CLINICAL TRIAL: NCT04680143
Title: Systemic Erythropoietin Injection in Patients Having Optic Atrophy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Fahmy Doheim, Prinicipal investigator, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0304845
Record Dates: First submitted 2020-12-15; First posted 2020-12-22 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Optic Atrophy
MeSH Terms: conditions — Optic Atrophy

STUDY DESIGN:
Intervention Model Description: The study included 10 patients diagnosed as post papilledemic optic atrophy that were attending Alexandria main university hospital. All patients underwent initially assessment of visual acuity, color vision, pupil reaction ,funduscopy and electrophysiological tests ( pattern visual evoked potential and pattern electroretinogram in both eyes to use data of the normal fellow eye as patients' internal control). Systemic erythropoietin injections (eprax 10000 IU subcutaneous twice daily for three days). Follow up after one month and three months by recording visual acuity and electro physiological studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systemic erythropoietin injections (Experimental): The study included 10 patients diagnosed as post papilledemic optic atrophy
  Interventions: Drug: Systemic erythropoietin injection

INTERVENTIONS:
Drug: Systemic erythropoietin injection — Systemic erythropoietin injections (eprax 10000 IU subcutaneous twice daily for three days).
  Other Names: Eprax 10000

SUMMARY:
The purpose of this treatment trial is to study the effect of systemic erythropoietin in patients having optic atrophy.

DETAILED DESCRIPTION:
The purpose of this treatment trial is to study the effect of systemic erythropoietin in patients having optic atrophy. The intervention is systemic erythropoietin injections (eprax 10000 IU subcutaneous twice daily for three days).

Follow up after one month and three months by recording visual acuity and electro physiological studies.

ELIGIBILITY:
Inclusion Criteria:

* Post papilledemic optic atrophy patients

Exclusion Criteria:

* Refuse to give an informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 3 months
  VIsual acuity assessed at the follow up
Pattern visual evoked Potential . | 3 months
  Pattern visual evoked Potential .in both eyes to use data of the normal fellow eye as patients' internal control
Pattern electroretinogram | 3 months
  Pattern electroretinogram in both eyes to use data of the normal fellow eye as patients' internal control

CONTACTS AND LOCATIONS:
Overall Officials: Mai ElBahwash, PhD, Principal Investigator — Alexandria Faculty of Medicine
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No